CLINICAL TRIAL: NCT04361734
Title: Understanding the Role Played by Serum and Membrane Lipids in Immune Cell Function in Patients With Systemic Lupus Erythematosus (SLE) and Healthy Donors
Brief Title: The Role of Lipids in Immune Cell Function in SLE Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: 15/0743
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — DNA; RNA; High-Energy Shock Waves; Nitroglycerin; Organization and Administration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Juvenile onset Systemic Lupus Erythematosus (SLE) patients: All patients who meet the American College of Rheumatology revised criteria for SLE who were diagnosed with SLE between the ages of 11 and 21.
  Interventions: Other: Blood sampling to include Deoxyribonucleic Acid (DNA) and Ribonucleic Acid (RNA)
- Adult onset Systemic Lupus Erythematosus (SLE) patients: All patients who meet the American College of Rheumatology revised criteria for SLE who were diagnosed with SLE between the ages of 24 and 80
  Interventions: Other: Blood sampling to include Deoxyribonucleic Acid (DNA) and Ribonucleic Acid (RNA)
- Matching healthy volunteers: Healthy volunteers, matched by age and gender, will be used as a control group
  Interventions: Other: Blood sampling to include Deoxyribonucleic Acid (DNA) and Ribonucleic Acid (RNA)

INTERVENTIONS:
Other: Blood sampling to include Deoxyribonucleic Acid (DNA) and Ribonucleic Acid (RNA) — * Blood sampling to measure immune cell phenotypes and examine DNA/RNA and identify serum biomarkers.
  * Food Frequency Questionnaires (FFQs) and/or diet recall questionnaires to assess dietary intake.
  * Cardiovascular Ultrasound Scans (USS) to measure how well blood is carried around the body.
  Other Names: Food Frequency Questionnaires (FFQs) and/or 24 hour diet recall questionnaires; Ultrasound Scan (USS); GTN (glyceryl trinitrate) administration

SUMMARY:
The overall aim of this project is to investigate the different types of immune cells found in the blood of patients with Systemic Lupus Erythematosus (SLE) and healthy donors. We know that the amount of fat on the surface of immune cells is an important factor controlling their behaviour. Immune cells from SLE patients are defective and this is associated with changes in the levels of fat on these cells. This project will investigate the level of fat in the blood and on immune cells from patients with SLE and age matched healthy controls, and measure how changes in the amount of fat can affect the way immune cells behave.

DETAILED DESCRIPTION:
Accelerated atherosclerosis is a serious complication of autoimmunity including patients with both adult and juvenile onset systemic lupus erythematosus (SLE). This suggests that defects in fat levels could contribute to disease pathogenesis. The immune system in patients with SLE does not work normally. In adult patients with SLE we know that many of the immune cells involved in protecting the body from infections or cancer are over-active and actually cause disease. In young people the immune system is still developing and very little is known about what goes wrong in patients that develop juvenile-onset SLE, whether this is the same as adult disease and whether the same treatments are relevant for this group of patients. This project aims to find out whether immune cells from SLE patients with adult-onset disease have the same defects as adult patients with juvenile-onset SLE. We know that an important factor that controls immune cell behaviour is the amount of fat that they have on their surface. We also know that a change in fat on immune cells from adult patients with SLE makes them defective. This project will investigate the level of fat in the blood and in immune cells from adult patients with juvenile-onset SLE and age matched healthy controls, and measure how changes in the amount of fat can affect the way immune cells behave. We will investigate how drugs that control fat levels can help to normalize the behaviour of immune cells from SLE patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE according to American College of Rheumatology revised criteria
* Having given written informed consent prior to undertaking any study-related procedures.
* Male and female patients between the ages of 18 and 80 years.

Patients who have met all the above inclusion criteria listed and healthy donors will be screened for the following exclusion criteria:

Exclusion Criteria:

* Under any administrative or legal supervision.
* Conditions/situations such as:
* A concomitant autoimmune disease
* Impossibility to meet specific protocol requirements (e.g. blood sampling).
* Patient is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.
* Uncooperative or any condition that could make the patient potentially non-compliant to the study procedures.
* Pregnant or breast-feeding women, currently or in the last three months prior to inclusion.
* Patients who have been vaccinated in the last three months prior to inclusion.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be approached by the consultant rheumatologist when the patient is attending their normal outpatient clinic appointment.
  Healthy donors will be approached in a similar way using information flyers, invitation letters and participant information sheets by a member of the research team.
  Healthy volunteers from UCL staff will be made aware of the study and also asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-02-15 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Collection of blood samples | 4 hours from point of sample collection
  Blood sampling to measure immune cell phenotypes and examine DNA/RNA and identify serum biomarkers.
Completion of FFQ's and/or diet recall questionnaires | Same day as recruited to study.
  FFQ's and/or diet recall questionnaires to assess dietary intake
Cardiovascular Ultrasound scans (USS) | Within 2 months from recruitment.
  USS of Intima Media Thickness (IMT), Flow Mediated Dilatation (FMD), Pulse Wave Velocity (PWV) and Laser Doppler Flowmetry measurement. As part of the procedure, sub lingual administration of GTN spray will be administered to measure FMD.

CONTACTS AND LOCATIONS:
Overall Officials: David Isenberg, Prof, Principal Investigator — UCL & University College London Hospitals NHS Foundation Trust
Locations (1):
- University College London Hospitals NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
All participants are required to indicate in written consent if they agree to the use of any left over samples and associated data for future research use.